CLINICAL TRIAL: NCT01218386
Title: Programmation of GnRH Antagonist Cycles With Estradiol Valerate: Impact on the Stimulation in IVF/ICSI.
Brief Title: Pretreatment With Estradiol Valerate
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Universitair Ziekenhuis Brussel (Other)
Responsible Party: Principal Investigator, Blockeel Christophe, Dr, Universitair Ziekenhuis Brussel
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2010-019924-30
Record Dates: First submitted 2010-10-08; First posted 2010-10-11 (Estimated); Last update posted 2012-03-28 (Estimated); Status verified 2012-03

CONDITIONS: Infertility
Keywords: ICSI; GnRH antagonists; planning
MeSH Terms: conditions — Infertility | interventions — Estradiol

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Study Group (Experimental): Start with estradiol valerate (Progynova, 2x2mg per day, 2mg in the morning, 2mg in the evening), orally, during 6-10 consecutive days from day 25 of the cycle onwards.
  If day 25 is Monday: 6 days Tuesday: 10 days Wednesday: 9 days Thursday: 8 days Friday: 7 days Saturday: 6 days Sunday: 6 days of Progynova, 2x2 mg per day After this pretreatment: Standard GnRH antagonist treatment protocol with start rFSH (Puregon®) at a dose of 150 IU From day 2 of the cycle onwards; GnRH antagonist (Orgalutran®) initiation on D6 of the stimulation
  Interventions: Drug: Estradiol valerate
- Control group (Active Comparator): Standard GnRH antagonist treatment protocol with start rFSH (Puregon®) at a dose of 150 IU From day 2 of the cycle onwards; GnRH antagonist (Orgalutran®) initiation on D6 of the stimulation
  Interventions: Drug: Estradiol valerate

INTERVENTIONS:
Drug: Estradiol valerate — Experimental group: estradiol valerate (Progynova, 2x2mg per day, 2mg in the morning, 2mg in the evening), orally, during 6-10 consecutive days from day 25 of the cycle onwards.
  Both groups:start rFSH (Puregon®) at a dose of 150 IU GnRH antagonist (Orgalutran®) initiation on D6 of the stimulation.
  Other Names: Progynova

SUMMARY:
The present study is set up to evaluate the efficacy of a programmation by administration of estrogen valerate during 6 or more consecutive days. In this prospective randomised trial, we study the impact of administration of Progynova® during 6, 7,8 9 or 10 consecutive days during the luteo-follicular transition period of the menstrual cycle.

DETAILED DESCRIPTION:
See Section Interventions

ELIGIBILITY:
Inclusion Criteria:

< 36 years old on day of randomisation FSH < 12 (in the early follicular phase) Normal ultrasound scan, i.e. presence of both ovaries, without evidence of abnormality within 6 months prior to randomisation.

Regular menstrual cycles of 21-35 days, presumed to be ovulatory. BMI between 18 and 29 (both inclusive) 1st or 2nd trial IVF or ICSI

Exclusion Criteria:

≥ 36 years old on day of randomisation Endometriosis ≥ grade 3 PCOS Poor responders (development of < 4 follicles in a previous IVF/ICSI cycle) Endocrine or metabolic abnormalities (pituitary, adrenal, pancreas, liver or kidney)

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 2010-05; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
number of egg retrievals on weekend days | up to 9 months

SECONDARY OUTCOMES:
The mean number of coc in each treatment group | up to 9 months

CONTACTS AND LOCATIONS:
Overall Officials: Paul Devroey, MD, PhD, Study Director — Universitair Ziekenhuis Brussel
Locations (1):
- UZ Brussel, Centre for Reproductive Medicine, Brussels, Belgium